CLINICAL TRIAL: NCT01872351
Title: Assessment of Chronic Fatigue Syndrome as a Mitochondrial Disorder
Brief Title: Therapy for Chronic Fatigue Syndrome: A Presumptive Mitochondrial Disorder
Status: Withdrawn | Type: Observational
Why Stopped: PI left the institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAI1410
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Fatigue Syndrome
Keywords: chronic fatigue syndrome; mitochondrial disorder; conditioning exercise; nutraceutical supplements; high protein diet
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Mitochondrial Diseases | interventions — Dietary Supplements; Acetylcarnitine; BID protein, human; Thioctic Acid; coenzyme Q10; Geritol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pre and 12 months post ENT: Compare the clinical status of CFS patients after at least 12 months of ENT to their status before ENT.
  ENT consists of:
  Daily conditioning exercise: 35-40 minutes
  Nutraceutical supplements: acetyl-L-carnitine 500 mg bid, alpha-lipoic acid (Alpha Lipoic Sustain 300) 300 mg qd, CoQ10 (Ubiquinol QH-absorb) 100 mg qd, docosahexanoic acid (maxDHA) 300 mg qd, plus a multivitamin (Centrum Silver) ½ tab bid.
  Diet: 25% protein, 35- 40% carbohydrate, 35-40% fat
  Interventions: Drug: Nutraceuticals

INTERVENTIONS:
Drug: Nutraceuticals
  Other Names: Jarrow Formulas:; - acetyl-L-carnitine 500 mg bid; - alpha-lipoic acid (Alpha Lipoic Sustain 300) 300 mg qd; - CoQ10 (Ubiquinol QH-absorb) 100 mg qd; - docosahexanoic acid (maxDHA) 300 mg qd; Pfizer Consumer Healthcare:; - multivitamin (Centrum Silver) ½ tab bid

SUMMARY:
The purpose of this study is to determine whether therapy that has been shown to be beneficial for mitochondrial diseases is also beneficial for Chronic Fatigue Syndrome (CFS) patients. This study is a chart review of previous CFS patients who received daily conditioning exercise, a high protein diet and nutraceutical therapy (ENT). Prescribed nutraceutical supplements included alpha-lipoic acid, acetyl-L-carnitine, omega-3fatty acids (maxDHA), coenzyme Q10 (CoQ10), plus a multivitamin.

Twelve CFS male and female patients between the ages of 20-70 years will be recruited to participate in this pilot study. Subjects will be eligible to participate if they meet the criteria for CFS of the Centers for Disease Control and Prevention (CDC). These include persistent, unexplained fatigue for at least 6 months, concurrent with four of the following: impaired memory/concentration, sore throat, new headaches, unrefreshing sleep, muscle pain, multi-joint pain, tender lymph nodes, and post-exertional malaise.

DETAILED DESCRIPTION:
The etiology and pathogenesis of chronic fatigue syndrome (CFS) is poorly understood. Although therapies have been proposed, none has been particularly effective. A preceding viral infection is believed to cause mitochondrial dysfunction in genetically susceptible individuals, resulting in overwhelming fatigue, myalgia and brain fuzziness. The purpose of this study was to determine whether therapy that has been shown to be beneficial for mitochondrial diseases is also beneficial for CFS.

Patients received daily conditioning exercise, a high protein diet and nutraceutical therapy (ENT). Prescribed nutraceutical supplements incldued alpha-lipoic acid, acetyl-L-carnitine, omega-3fatty acids (maxDHA), coenzyme Q10 (CoQ10), plus a multivitamin, which were selected to enhance mitochondrial function and antioxidant action. Following the institution of ENT, patients had received this therapy for varying lengths of time, ranging from 12 to 40 months.

ELIGIBILITY:
Inclusion Criteria:

Severe chronic fatigue for 6 or more consecutive months 4 or more of the following 8 symptoms concurrently:

* post-exertion malaise lasting more than 24 hours
* unrefreshing sleep
* significant impairment of short-term memory or concentration
* muscle pain
* pain in the joints without swelling or redness
* headaches of a new type, pattern, or severity
* tender lymph nodes in the neck or armpit
* a sore throat that is frequent or recurring These symptoms should have persisted or recurred during 6 or more consecutive months of illness and they cannot have first appeared before the fatigue.

Exclusion Criteria:

* Additional medical illnesses causing chronic fatigue
* Ongoing exertion

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twelve CFS male and female patients between the ages of 20-70 years will be recruited to participate in this pilot study. Subjects will be eligible to participate if they meet the criteria for CFS of the Centers for Disease Control and Prevention (CDC). These include persistent, unexplained fatigue for at least 6 months, concurrent with four of the following: impaired memory/concentration, sore throat, new headaches, unrefreshing sleep, muscle pain, multi-joint pain, tender lymph nodes, and post-exertional malaise. Subjects will be screened for eligibility; the study will be explained and a verbal consent will be given over the telephone. If the subject agrees, they will be sent a questionnaire assessing their clinical and fatigue status prior to starting ENT and their present clinical and fatigue status, as well as their compliance to ENT.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Modified Fatigue Severity Score (FSS-11) | 6-40 months

SECONDARY OUTCOMES:
Other Symptoms Questionnaire score | 6-40 months
  Assess pre/post symptoms of CFS not covered by the Modified Fatigue Severity Score

OTHER OUTCOMES:
Compliance Questionnaire score | First 6 months vs. last 6 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Slonim, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States